CLINICAL TRIAL: NCT05010395
Title: Increasing Health Insurance Enrollment Among Uninsured Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Office of Evaluation Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Yokum, Director of The Policy Lab, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 02152015
Record Dates: First submitted 2021-07-09; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Health Behavior
Keywords: health insurance enrollment
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Control (No Intervention): Individuals in this arm did not receive a letter.
- Arm 1: Basic Letter (Experimental): Individuals received a letter with information about the benefits of enrolling, the February 15th sign-up deadline, the HealthCare.gov website, and the call center phone number.
  Interventions: Behavioral: Letter intervention
- Arm 2: Action (Experimental): Individuals in this arm received a letter that emphasized only minimal marginal effort is required; and used adjectives and verbs connoting action (e.g., "almost done," "quick," "act now," and "fast").
  Interventions: Behavioral: Letter intervention
- Arm 3: Action, Implementation (Experimental): Individuals in this arm received a letter similar to Arm 2, but with the addition of a calendar that draws attention to the February 15th deadline; and provided fill-in blanks in which the recipient can write the planned month, day, and time when they intend to enroll.
  Interventions: Behavioral: Letter intervention
- Arm 4: Action, Implementation, Picture (Experimental): Individuals in this arm received a letter similar to Arms 2 and 3, but with the addition of an image of then HealthCare.gov Chief Executive Officer Kevin Counihan
  Interventions: Behavioral: Letter intervention
- Arm 5: Norm (Experimental): Individuals in this arm received a letter that included the following social norm sentence: "Americans are enrolling but you haven't joined them."
  Interventions: Behavioral: Letter intervention
- Arm 6: Norm, Pledge (Experimental): Individuals in this arm received a letter that included a statement, to be checked in agreement, that "I pledge to Get Covered at Healthcare.gov."
  Interventions: Behavioral: Letter intervention
- Arm 7: Loss Aversion (Experimental): Individuals in this arm received a letter that warned "You risk paying a fee of $325 or 2% of your income-whichever is higher."
  Interventions: Behavioral: Letter intervention
- Arm 8: Kitchen Sink (Experimental): Individuals in this arm received a letter that includes all behavioral dynamics except for the pledge (due to space limitations).
  Interventions: Behavioral: Letter intervention

INTERVENTIONS:
Behavioral: Letter intervention — Letter intervention
  Arms: Arm 1: Basic Letter; Arm 2: Action; Arm 3: Action, Implementation; Arm 4: Action, Implementation, Picture; Arm 5: Norm; Arm 6: Norm, Pledge; Arm 7: Loss Aversion; Arm 8: Kitchen Sink

SUMMARY:
This randomized evaluation used behaviorally-informed letters to increase health insurance take-up on the Affordable Care Act (ACA) Marketplaces.

DETAILED DESCRIPTION:
During Open Enrollment Periods for the ACA Marketplaces, qualifying individuals can purchase health insurance plans through the Federal Health Insurance Marketplace (FHIM). As of early February 2015, many people had visited HealthCare.gov and started an online account, but not yet selected a plan. The Department of Health and Human Services (HHS), in collaboration with the Office of Evaluation Sciences (OES), developed and sent letters to assist these individuals with completing their enrollment before the deadline.

To evaluate the effect of the letters, the team used a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Those with an English language preference; those who had not enrolled in an ACA plan as of early February 2015

Exclusion Criteria:

* Those with a Spanish language preference

This intervention was a program evaluation and did not go through Human Subjects Protection Review.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 811795 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2015-02-15 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Percent of individuals enrolling in an ACA plan by the end of the Open Enrollment period. | Two weeks
  Percent of individuals enrolling in an ACA plan during the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: David Yokum, PhD, Principal Investigator — Brown University

IPD SHARING:
Plan to Share IPD: Yes
Deidentified replication data will be posted to OSF upon manuscript acceptance.
Supporting Information: Study Protocol, Analytic Code
URL: https://osf.io/pb256/

REFERENCES:
- [Derived] Yokum D, Hopkins DJ, Feher A, Safran E, Peck J. Effectiveness of Behaviorally Informed Letters on Health Insurance Marketplace Enrollment: A Randomized Clinical Trial. JAMA Health Forum. 2022 Mar 4;3(3):e220034. doi: 10.1001/jamahealthforum.2022.0034. eCollection 2022 Mar. PMID 35977283